CLINICAL TRIAL: NCT00574067
Title: Buprenorphine for Prisoners
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01DA021579-01A1 (NIH); R01DA021579 (NIH); 1R01DA021579-01A1 (NIH)
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Heroin Addiction
MeSH Terms: conditions — Heroin Dependence | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Buprenorphine+OTP (Experimental): Buprenorphine and counseling in prison and continued at opioid treatment program (OTP) upon release.
  Interventions: Drug: Buprenorphine +OTP
- Buprenorphine+CHC (Experimental): Buprenorphine and counseling in prison and continued at a community health center (CHC) upon release.
  Interventions: Drug: Buprenorphine +CHC
- Counseling + OTP (Active Comparator): Counseling only in prison and Buprenorphine upon release at a opioid treatment program (OTP)
  Interventions: Drug: Counseling +OTP
- Counseling + CHC (Active Comparator): Counseling only in prisons and Buprenorphine upon release at a community health center (CHC)
  Interventions: Drug: Counseling +CHC

INTERVENTIONS:
Drug: Buprenorphine +OTP — Buprenorphine thrice weekly and counseling for four months while in pre-release prison, with referral for continued treatment at an opioid agonist treatment (OTP) program upon release. Such treatment lasts for 1 year in the community. Buprenorphine dosage, following an induction period,is 32 mg Mondays and Wednesdays and 48 mg Fridays
  Other Names: Suboxone
  Arms: Buprenorphine+OTP
Drug: Buprenorphine +CHC — Buprenorphine thrice weekly and counseling provided in pre-release prison for 4 months, with referral for continued treatment for 1 year in the community at a community health center (CHC). Following an induction period, buprenorphine dosing will be 32 mg on Mondays and Wednesdays and 48 mg on Fridays.
  Other Names: Suboxone
  Arms: Buprenorphine+CHC
Drug: Counseling +OTP — Counseling only for 4 months in pre-release prison, with referral upon release for buprenorphine treatment and counseling at an opioid agonist treatment program to last for 1 year. Following an induction period, buprenorphine dosing will be thrice weekly, with 32 mg on Mondays and Wednesdays and 48 mg on Fridays.
  Other Names: Suboxone
  Arms: Counseling + OTP
Drug: Counseling +CHC — Counseling only for 4 months in pre-release prison, with referral upon release for buprenorphine treatment and counseling at a community health center to last for 1 year. Following an induction period, buprenorphine dosing will be thrice weekly, with 32 mg on Mondays and Wednesdays and 48 mg on Fridays.
  Other Names: Suboxone
  Arms: Counseling + CHC

SUMMARY:
This five-year study examines the effectiveness of buprenorphine treatment provided to previously-addicted inmates(N=320; 160 males, 160 females) initiated in prison and continued in the community. The study also examines the extent to which the setting of post-release buprenorphine is provided.It is expected that participants receiving in-prison buprenorphine will have superior outcomes compared to participants who did not receive in-prison buprenorphine.

DETAILED DESCRIPTION:
Participants will be randomly assigned, within gender, to one of four treatment conditions: 1) buprenorphine and counseling in prison, with referral for continued treatment at an OTP upon release; 2) buprenorphine and counseling in prison, with referral for continued treatment at a CHC upon release; 3) counseling only in prison, with referral for buprenorphine and counseling at a OTP upon release; and 4) counseling only in prison, with referral for buprenorphine and counseling at a CHC upon release. Participants will be assessed at study entry and at 1, 3, 6, and 12 months following their release from prison. Outcome measures include: treatment entry and retention in the community, heroin use, cocaine use, HIV infection, HIV-risk behaviors, criminal activity, and employment.

ELIGIBILITY:
Inclusion Criteria:

1. pre-release prison inmate with 3-6 months remaining until planned release
2. history of heroin dependence(meeting DSM-IV criteria of heroin dependence at the time of incarceration and manifesting physical dependence during the year preceding incarceration
3. suitability for buprenorphine treatment as determined by medical evaluation
4. willingness to participate in the study
5. having a Baltimore address and planning to live in Baltimore after release from prison -

Exclusion Criteria:

1. evidence of kidney failure
2. evidence of liver failure
3. history of psychosis
4. having a pending parole hearing
5. unadjudicated charges that could result in additional prison time or transfer to another facility -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 213 (Actual)
Dates: Start 2008-09; Primary Completion 2013-03 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Metropolitan Transition Center, Baltimore, Maryland
  - Maryland Correctional Institution for Women, Jessup, Maryland

REFERENCES:
- [Background] Kinlock TW, Gordon MS, Schwartz RP, Fitzgerald TT. Developing and Implementing a New Prison-Based Buprenorphine Treatment Program. J Offender Rehabil. 2010 Feb;49(2):91-109. doi: 10.1080/10509670903534951. PMID 20473351
- [Background] Gordon MS, Kinlock TW, Schwartz RP, Couvillion KA, O'Grady KE. The Severity, Frequency, and Variety of Crime in Heroin-Dependent Prisoners Enrolled in a Buprenorphine Clinical Trial. Prison J. 2013 Dec 1;93(4):390-410. doi: 10.1177/0032885513500753. PMID 25392564
- [Derived] Blue TR, Gordon MS, Schwartz RP, Couvillion K, Vocci FJ, Fitzgerald TT, O'Grady KE. Longitudinal analysis of HIV-risk behaviors of participants in a randomized trial of prison-initiated buprenorphine. Addict Sci Clin Pract. 2019 Dec 2;14(1):45. doi: 10.1186/s13722-019-0172-2. PMID 31787108

RESULTS

PARTICIPANT FLOW:
Groups:
- Bup+OTP: Buprenorphine: Buprenorphine thrice weekly and counseling for four months while in pre-release prison, with referral for continued treatment at an opioid agonist treatment program upon release. Such treatment lasts for 1 year in the community. Buprenorphine dosage, following an induction period,is 32 mg Mondays and Wednesdays and 48 mg Fridays
- Bup+CHC: Buprenorphine: Buprenorphine thrice weekly and counseling provided in pre-release prison for 4 months, with referral for continued treatment for 1 year in the community at a community health center. Following an induction period, buprenorphine dosing will be 32 mg on Mondays and Wednesdays and 48 mg on Fridays.
- Counseling+OTP: Buprenorphine: Counseling only for 4 months in pre-release prison, with referral upon release for buprenorphine treatment and counseling at an opioid agonist treatment program to last for 1 year. Following an induction period, buprenorphine dosing will be thrice weekly, with 32 mg on Mondays and Wednesdays and 48 mg on Fridays.
- Counseling+CHC: Buprenorphine: Counseling only for 4 months in pre-release prison, with referral upon release for buprenorphine treatment and counseling at a community health center to last for 1 year. Following an induction period, buprenorphine dosing will be thrice weekly, with 32 mg on Mondays and Wednesdays and 48 mg on Fridays.
Period: Overall Study
Arm/Group | Bup+OTP | Bup+CHC | Counseling+OTP | Counseling+CHC
Started | 53 | 53 | 54 | 53
Completed | 52 | 52 | 54 | 53
Not Completed | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- B+OTP: Buprenorphine: Buprenorphine thrice weekly and counseling for four months while in pre-release prison, with referral for continued treatment at an opioid agonist treatment program upon release. Such treatment lasts for 1 year in the community. Buprenorphine dosage, following an induction period,is 32 mg Mondays and Wednesdays and 48 mg Fridays
- B+CHC: Buprenorphine: Buprenorphine thrice weekly and counseling provided in pre-release prison for 4 months, with referral for continued treatment for 1 year in the community at a community health center. Following an induction period, buprenorphine dosing will be 32 mg on Mondays and Wednesdays and 48 mg on Fridays.
- C+OTP: Buprenorphine: Counseling only for 4 months in pre-release prison, with referral upon release for buprenorphine treatment and counseling at an opioid agonist treatment program to last for 1 year. Following an induction period, buprenorphine dosing will be thrice weekly, with 32 mg on Mondays and Wednesdays and 48 mg on Fridays.
- C+CHC: Buprenorphine: Counseling only for 4 months in pre-release prison, with referral upon release for buprenorphine treatment and counseling at a community health center to last for 1 year. Following an induction period, buprenorphine dosing will be thrice weekly, with 32 mg on Mondays and Wednesdays and 48 mg on Fridays.
- Total: Total of all reporting groups
Arm/Group | B+OTP | B+CHC | C+OTP | C+CHC | Total
Number analyzed (Participants) | 52 | 52 | 54 | 53 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.15 (7.5) | 39.18 (8.7) | 39.55 (10.0) | 38.42 (9.1) | 39.08 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 16 | 15 | 63
  Male | 37 | 35 | 38 | 38 | 148

OUTCOME MEASURES:

1. Primary Outcome: Number of Days of Heroin Use
Description: mean days used heroin during the past 30 days
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bup+OTP | Bup+CHC | Counseling+OTP | Counseling+CHC
Number analyzed (Participants) | 52 | 52 | 54 | 53
days | 6.0 (11.4) | 6.4 (11.5) | 6.5 (11.3) | 4.0 (9.0)

2. Primary Outcome: Drug Abuse Treatment Entry and Retention in the Community
Description: entered community treatment within 10 days of release from prison (yes vs. no)
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | B+OTP | B+CHC | C+OTP | C+CHC
Number analyzed (Participants) | 52 | 52 | 54 | 53
participants | 22 | 26 | 23 | 11

3. Secondary Outcome: Number of Days of Cocaine Use
Description: Number of days used cocaine during the past 30 days.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bup+OTP | Bup+CHC | Counseling+OTP | Counseling+CHC
Number analyzed (Participants) | 52 | 52 | 54 | 51
days | 1.1 (4.3) | 4.1 (9.5) | 4.7 (9.4) | 2.7 (6.0)

4. Secondary Outcome: Criminal Activity
Description: Days of crime during the past 30 days
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bup+OTP | Bup+CHC | Counseling+OTP | Counseling+CHC
Number analyzed (Participants) | 52 | 52 | 54 | 51
days | 3.4 (9.4) | 5.4 (11.4) | 3.3 (9.2) | 3.2 (9.0)

5. Secondary Outcome: Employment Status
Description: Number of days employed during the past year
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: days
Arm/Group | B+OTP | B+CHC | C+OTP | C+CHC
Number analyzed (Participants) | 52 | 52 | 54 | 53
days | 30.0 (28.1) | 29.6 (26.9) | 22.3 (32.4) | 31.4 (30.1)

6. Secondary Outcome: HIV Risk Behavior Needle Sharing
Description: Number of times shared a needle during the past year
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: times
Arm/Group | B+OTP | B+CHC | C+OTP | C+CHC
Number analyzed (Participants) | 52 | 52 | 54 | 53
times | 2.9 (15.9) | .1 (.5) | 2.1 (13.6) | .1 (1.3)

7. Secondary Outcome: HIV Risk Behavior
Description: Number of times had sex without using a condom during the past year
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: times
Arm/Group | B+OTP | B+CHC | C+OTP | C+CHC
Number analyzed (Participants) | 52 | 52 | 54 | 53
times | 59.7 (52.6) | 36.1 (40.3) | 33.3 (29.3) | 50.4 (38.4)

ADVERSE EVENTS:
Description: 0 represents other [non-serious] adverse events were not collected/assessed during the 12-months post-release time period.
Arm/Group | B+OTP | B+CHC | C+OTP | C+CHC
Serious Adverse Events (participants affected / at risk) | 4/52 | 14/52 | 10/54 | 10/53
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | B+OTP (N=52) | B+CHC (N=52) | C+OTP (N=54) | C+CHC (N=53)
constipation (Gastrointestinal disorders) | 1 (1) | 0/0 (0) | 0 (0) | 0 (0)
back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — fell off ladder.
swollen foot (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
unkown (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) — We were unable to obtain hospital medical records
depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
kidney problem (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
physical assualt (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
blood clot (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
alcohol withdrawal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
chest pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cesarean birth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
neck pain (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
shoulder pain (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pregnancy compplications (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
ulcer (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
allergic reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
gallstones (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
cellulitis in right arm and leg (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
osteomyelitis and soft tissue infection of the cervical spine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
seizure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pregnancy complications (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No